CLINICAL TRIAL: NCT05146427
Title: Pilot Study: Investigating Mood Changes After Slow-wave Enhancement
Acronym: SWE
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Equipment for slow wave enhancement is no longer available
Sponsor: University of Pennsylvania (Other)
Responsible Party: Principal Investigator, Philip Gehrman, Associate Professor, University of Pennsylvania
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 844797
Record Dates: First submitted 2021-11-11; First posted 2021-12-06 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Depressive Disorder, Major; Depression; Depression, Unipolar; Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major; Depression; Depressive Disorder

STUDY DESIGN:
Intervention Model Description: All participants will be randomized to active or sham enhancement for one week. For the second week, they will then receive the alternate condition.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Slow-wave enhancement (Experimental): Participants will wear the Philips SmartSleep Deep Sleep Headband which will play auditory tones to selectively enhance slow-wave activity.
  Interventions: Device: Slow-wave enhancement
- Sham Slow-wave enhancement (Sham Comparator): Participants will wear the Philips SmartSleep Deep Sleep Headband which will not be programmed to enhance slow-wave activity
  Interventions: Device: Sham device

INTERVENTIONS:
Device: Slow-wave enhancement — A headband that measures slow-wave activity during sleep and uses auditory stimulation to enhance slow waves using closed-loop auditory stimulation.
  Arms: Active Slow-wave enhancement
Device: Sham device — A headband that measures slow-wave activity during sleep but has no auditory stimulation.
  Arms: Sham Slow-wave enhancement

SUMMARY:
The aim of this pilot project proposal is to test the hypothesis that decreased sleep slow-wave activity (SWA) observed in individuals with major depressive disorder (MDD) is related to mood dysfunction, and that manipulating SWA may serve to improve mood by normalizing SWA regulation. The investigators propose to enhance SWA during nighttime sleep in a group of 20 antidepressant-free males and females age 25-50 with varying degrees of impairment in mood. Each participant will undergo one baseline night of sleep in the laboratory and then will sleep with the SmartSleep Headband nightly for two weeks in their own home. For one week, slow-wave sleep will be enhanced. On the alternate week, sleep will not be changed. Following the two weeks of sleeping with the device, participants will then spend another night in the sleep laboratory to assess changes in sleep. Mood will be assessed by self-report and clinician-administered scales following the baseline night of sleep, virtually after the first experimental week, and at the conclusion of the study.

ELIGIBILITY:
Inclusion Criteria:

1. Age 25-50 years.
2. Primary language is English.
3. Normal cognition.
4. Normal (or corrected-to-normal) vision and hearing.
5. Current depression.
6. Stable, normally-timed sleep-wake cycle as determined by interview, 1-week daily sleep log, and 1-week wrist actigraphic evidence, and defined by:

   1. Habitual nocturnal sleep duration between 6h and 9h.
   2. Habitual bedtime between 9pm-12am.
   3. No evidence of habitual napping.

Exclusion Criteria:

1. Current or prior medical condition that could interfere with collection or interpretation of data, based on medical history.
2. History of stroke, epilepsy, brain scarring, or head injury causing unconsciousness.
3. Independent/Intrinsic sleep disorder other than insomnia based on history or polysomnogram.
4. Recent use of psychoactive medications or medication thought to impact sleep or CNS function, as determined by investigators (e.g. SSRIs, benzodiazepines, glutamate modulators, gabapentin).
5. History of or current psychiatric conditions that increase study risk or grossly impair CNS function (e.g., current anorexia or bulimia, history of substance dependence or current substance abuse, lifetime history of psychosis).
6. Lifetime history of electroconvulsive therapy.
7. Pregnancy as determined by self-report.
8. Travel beyond 2 time zones in the 2 months before study.
9. Unwillingness to refrain from using alcohol or caffeine during the study.

Ages: 25 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in Quick Inventory of Depressive Symptoms | daily, up to 14 days
  Depression severity measure, score ranges from 0-27, higher scores indicate worse depressive symptoms

SECONDARY OUTCOMES:
Change from baseline in Visual Analog Scale - Mood | daily, up to 14 days
  measure of positive and negative mood, scores range from 0 to 100, higher scores indicate worse depressive symptoms
Change from baseline in Profile of Mood States | daily, up to 14 days
  measure of total mood disturbance, scores range from 0 to 28, higher scores indicate worse depressive symptoms
Change from baseline in Positive and Negative Affect Schedule | daily, up to 14 days
  measure of positive and negative affect, scores range from 10 to 50, higher scores indicate worse depressive symptoms

IPD SHARING:
Plan to Share IPD: No